CLINICAL TRIAL: NCT05923307
Title: Multifactorial Approach to Dementia. Multicentric Study
Brief Title: Multifactorial Approach to Dementia, Multicentric Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Daniel Serrani Azcurra (Other)
Collaborators: Zarebski Graciela, Kabanchik Alicia, Marconi Araceli (Unknown)
Responsible Party: Sponsor-Investigator, Daniel Serrani Azcurra, Principal researcher, Universidad Atlantida
Organization: Universidad Atlantida (Other)
Other Study IDs: 01569
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Dementia of Alzheimer Type; Dementia Frontotemporal; Narcissistic Personality Disorder; Depression; Personality Change
MeSH Terms: conditions — Pick Disease of the Brain; Narcissistic Personality Disorder; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess the role of narcisistic personality disorder and life stressful events in conversion rate to dementia, using a three tier approach along three research lines employing subjects with dementia in retrospective assessment, and normal subjects no yet developing demetia in prospective follow up. The main question[s] it aims to answer are:

* narcisistic personality disorder as risk factor for conversion to dementia
* life stressful events as risk factor for conversion to dementia Participants will be assessed with a complete neurocognitive battery, brain images studies, laboratory analysis, and sociodemographic profile, including depression and comorbidities.

DETAILED DESCRIPTION:
Previous studies have identified multiple risk factors for dementia in a variety of settings. However personality traits have received less attention as a contributing or mediating factor. The identification of potentially modifiable risk factors has been critical in the development of effective multifactorial intervention programmes for people at risk of dementia. Studies that examined the role of personality traits as risk factor for dementia recruited participants with mild cognitive impairment or mild to moderate dementia living in institutional or community settings. In this 3 tiered study, 3 lines of research will be pursued. In lines 1 and 2 retrospective analysis of patients with dementia will be performed searching for the mediating or predisposing role of narcissistic personality disorder as a risk factor for the development of dementia. in the 3rd line of research normal participants will complete a multifactorial baseline assessment of putative predictors of mild cognitive impairment or dementia and then will complete prospective cognitive, affective and personality diaries for a period of 12 months, in order to detect association of personality traits to dementia conversion.

Methods Ethics statement This study will be submitted to Ethics Committee of INICIEN Research Authority, and participants will be requested to give written informed consent in accordance with the declaration of Helsinki.

Design Longitudinal prospective and retrospective cohort study. Participant recruitment 3 lines of research. In line 1 and 2 patients with dementia will be assessed in a retrospective approach and in the line 3 healthy cases without cognitive impairment will be recruited to determine if narcisistic personality play a role in the risk of dementia onset (AD, frontotemporal dementia). Patients files and subjects will be recruited from multicenter Neurology, Old Age Psychiatry and Geriatric Medical secondary care outpatient clinics. Cases should be referred to these clinics for assessment, diagnosis and management by their primary care physician, or referred to a Psychiatrist by their clinical physician.

Inclusion and exclusion criteria All participants should be over 50 years of age in research line 1, and no age limit will be assumed for cases in reesarch lines 1 and 2. All diagnoses of dementia will be made according to DSM V criteria. Significant medical causes of dementia should be excluded during diagnostic investigations. Diagnoses will be made by operationalised criteria for dementia validated against neuropathological diagnosis Participants were excluded if they declined participation, died or withdrew from the study before commencing follow up period, unable to perform the assessments due to other co-morbid conditions, or were too visually impaired to complete cognitive assessments. Baseline Clinical Assessment All participants received a detailed baseline assessment to quantify putative risk factors for dementia. The factors included were selected on the basis of their previous identification as risk factors in more than one high quality study in older people, and/or their relevance to clinical features of dementia postulated to be causative of neurocognive disorder conversion.

Assessments included medical history (residence, history of life stressful events, affective state, sociodemographic factors). Objective assessments included the cognitive battery, personality assessment with narcisistic personality disorder, Yesavage depression scale. Participants were assessed at baseline and during follow up period of one year.

Dementia specific scales were used to assess specific staging level and dementia specific type, depression, and behavioural and psychological symptoms of dementia.

Outcome Measures The primary outcome measure will be dementia conversion occurring during the 12 month follow up period. Secondary outcome measures will be proportional hazard ratios for time to dementia conversion, according to diagnosis and status of personality disorder narcisistic type as putative clinical predictor. If the participants did not show off at previously assigned points, they will be reminded by telephone after 2 weeks. The caregiver will be asked to assist in the completion of diaries when dementia is present.

Statistics Differences in baseline characteristics across groups will be compared using Fisher's Exact test for categorical data, ANOVA for normally distributed data and Kruskal-Wallis for non-normally distributed data. Differences between individual groups will be compared using the Chi squared test for categorical data, Student's t test for normally distributed data and Mann-Whitney U test for non-normally distributed data.

In case of censoring of data from some participants (as a result of death or withdrawal from the study), Cox regression (adjusted for age and sex) will be used to obtain a proportional hazard ratio for personality disorder as risk factor to dementia conversion. Loglinear Poisson regression models (adjusted for age and sex) will be used to obtain an incidence density ratio for dementia and its subtypes in comparison with healthy controls. without personality disorders In order to examine the associations between exposure to narcisitic personality disorder as risk factors for dementia conversion in those participants with dementia, Cox regression will be used to obtain univariate proportional hazard ratios for each risk factor, adjusted for age and sex, using time to the occurrence of at least mild cognitive impairment as the dependent variable. Hazard ratios will be given according to presence or absence of the risk factor, or per point on quantitative scales as appropriate. Analyses will be performed initially for all participants with or without dementia, and then repeated stratified by diagnosis.

Following identification in univariate models, significant and potentially modifiable risk factors will be entered into a multivariate forward stepwise Cox regression model, p 0.05 for entry, p 0.1 for removal. Age and sex will be included even if not significant. Where similar clinical features coould be described by more than one significant risk factor the factor with the higher level of significance in univariate analyses will be entered into multivariate analyses, in order to avoid co-aggregation of predictors.

ELIGIBILITY:
Inclusion Criteria:

research line 3

* healthy subjects over 50 years of age.
* diagnosis of dementia should be made according to DSM V criteria.
* Diagnoses made by operationalised criteria for dementia

Exclusion Criteria:

* Participants excluded if declined participation, died or withdrew from the study
* unable to perform the assessments due to other co-morbid conditions
* were too visually impaired to complete cognitive assessments.

in research lines 1 and 2 inclusion criteria subjects with confirmed diagnosis of dementia

* putative narcisistic personality disorder
* no age limit

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals eligible to participate were diagnosed with dementia, or had inconclusive results living at the community or residential institutions invited to attend a follow-up, cognitively healthy or minimally impaired, or had mild cognitive impairment (MCI), or dementia
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
new onset of dementia during the follow-up period | 1 year
  dementia diagnosed according to the Diagnostic and Statistical Manual of Mental Disorders V, considered affected by dementia when agreement on this diagnosis was reached between a psychologist and a geriatrician. If the physicians failed to agree, the diagnosis had to be confirmed by a second geriatrician.

SECONDARY OUTCOMES:
univariate proportional hazard ratios for narcissistic personality as risk factor, adjusted for age and sex | 1 year
  Hazard ratios are given according to presence or absence of the risk factor, or per point on quantitative scales as appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- universidad Atlantida, Buenos Aires, Outside U.S. and Canada, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fiest KM, Jette N, Roberts JI, Maxwell CJ, Smith EE, Black SE, Blaikie L, Cohen A, Day L, Holroyd-Leduc J, Kirk A, Pearson D, Pringsheim T, Venegas-Torres A, Hogan DB. The Prevalence and Incidence of Dementia: a Systematic Review and Meta-analysis. Can J Neurol Sci. 2016 Apr;43 Suppl 1:S3-S50. doi: 10.1017/cjn.2016.18. PMID 27307127
- [Result] Ganguli M, Dodge HH, Chen P, Belle S, DeKosky ST. Ten-year incidence of dementia in a rural elderly US community population: the MoVIES Project. Neurology. 2000 Mar 14;54(5):1109-16. doi: 10.1212/wnl.54.5.1109. PMID 10720283
- [Result] serrani daniel Narcissism Vulnerability as Risk Factor for Alzheimer´s Disease- A Prospective Study Austin J Clin Neurol 2015;2(7): 1057.
- [Result] Chatterjee A, Strauss ME, Smyth KA, Whitehouse PJ. Personality changes in Alzheimer's disease. Arch Neurol. 1992 May;49(5):486-91. doi: 10.1001/archneur.1992.00530290070014. PMID 1580810
- [Result] Wilson RS, Schneider JA, Arnold SE, Bienias JL, Bennett DA. Conscientiousness and the incidence of Alzheimer disease and mild cognitive impairment. Arch Gen Psychiatry. 2007 Oct;64(10):1204-12. doi: 10.1001/archpsyc.64.10.1204. PMID 17909133